CLINICAL TRIAL: NCT05540171
Title: An Educational Intervention Program to Improve the Oral Health of HIV-Positive Children in Kano, Nigeria.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aminu Kano Teaching Hospital (Other)
Collaborators: NIH Office of AIDS Research (OAR) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Yewande Isabella Adeyemo, Dr., Aminu Kano Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NHREC/17/03/2018; 2D43TW010543-06 (NIH)
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: HIV; Dental Caries; Quality of Life; Oral Disease; Oral Infection; Oral Manifestations
Keywords: HIV; Children; Oral Health Status; Oral Health Related Quality of Life; Kano; Self oral care; Oral health education; Randomized controlled study
MeSH Terms: conditions — Dental Caries; Mouth Diseases; Oral Manifestations | interventions — Health Education, Dental

STUDY DESIGN:
Intervention Model Description: A 2-arm randomized control study which involves two groups of participants who will be recruited into the study at the sites. The sites would have been randomized into control and intervention arms using a simple lottery technique.
  Four (4) identical slips of paper with 'control' printed on 2 on them and 'intervention' on the other 2 slips will be provided. Each paper will be sealed in envelopes which will all be identical, and they will be placed in a box. An individual unconnected to the study will be asked to select two (2) envelopes from the box and these will be assigned the control group while the two (2) envelopes left in the box will be the assigned the intervention group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistants (dentists) collecting data and the study statistician will be blinded as to which sites are the intervention and control arms.
  The primary investigator and instructor will not be blinded as knowledge of the intervention will be necessary to ensure proper implementation of the intervention protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education intervention (Oral health education and instructions/training for self-oral care) (Experimental): The intervention arm will be given a 45 minute oral health education which will include oral hygiene instructions and motivation/training for oral self-care (dietary counselling; snacking during and not mealtimes; post-meal rinsing; flossing; brushing frequency, time, and method; tongue cleaning; toothbrush type/care; toothpaste quantity/type; dental visits). Audio-visual aids and leaflets reinforcing the oral health education will also be provided.
  Interventions: Other: Oral health education and instructions/training for self-oral care
- No intervention (Control) (No Intervention): The control arm/group will receive no intervention (Oral health education) until right after the study is over.

INTERVENTIONS:
Other: Oral health education and instructions/training for self-oral care — Education intervention
  Arms: Education intervention (Oral health education and instructions/training for self-oral care)

SUMMARY:
The aim of this 2- arm randomized-control study is to determine the effect of an oral hygiene self care intervention on the oral health status and oral health-related quality of life (OHRQoL) of HIV-positive children (age: 8-16 years, n=172) presenting to five pediatric HIV clinics in Kano, Nigeria.

The intervention will comprise oral health education and instructions on oral self-care.

Data on oral health status and OHRQoL will be obtained at baseline and at 1, 3 and 6 months.

Study findings will help inform policies to improve the oral health and OHRQoL of HIV-positive Nigerian children and guide the integration of oral health care services into HIV programs.

DETAILED DESCRIPTION:
The paediatric HIV clinic sites will be randomized into intervention and control groups and all consecutive consenting eligible participants will be recruited and enrolled into the study at the sites until the estimated sample size for each study arm (86 participants per arm) is reached. The number of participants per arm will be allocated in proportions observed from each site's population. Baseline data collection will commence after all participants have been screened, recruited, and enrolled. The intervention arm will consist of oral health education and demonstration of how to perform oral self-care.

Hypothesis: There will be a mean difference of 0.5 in children's oral hygiene scores between intervention and control arms at 6 months post-intervention.

Based on reported oral hygiene score standard deviation=0.96, desired power=0.90, Type I error rate=0.05, we need 77 participants/arm to detect a clinically meaningful mean difference of 0.5 in oral hygiene score between intervention and control arms at 6 months post-intervention.

To account for possible loss to follow-up over 6 months, the participants' total sample size was increased to 172 (86 participants/arm).

Ethical Approval: Has been obtained from Aminu Kano Teaching Hospital (AKTH) and Kano State research ethics committees.

Study instrument/measures:

1. Socio-demographic/clinical information: Age, gender, family size, household income, caregiver occupation/education, birth order/rank, HIV status of caregiver (self-reported/extracted from records), child's antiretroviral treatment (ART) regimen, comorbidities, most recent viral load, helper T cells (CD4+) count.
2. OHRQoL: The child perception questionnaire (CPQ) captures global ratings of child's oral health; four domains: oral symptoms, functional limitations, emotional and social well-being; Likert scale ('never'=0 to everyday/ almost every day'=4). The questionnaire will be translated into Hausa.
3. Oral health status:

   i. Decayed, Missing, and Filled Teeth (DMFT/dmft) index, scored: D/d, M/m, F/f.

   ii. International Caries Detection and Assessment System, (ICDAS) (caries severity) (0=sound tooth- 6=distinctly cavitated tooth).

   iii. Pulp (visible), Ulceration (oral mucosa), Fistula and Abscess due to caries (PUFA/pufa) index scored: P/p, U/u, F/f, A/a.

   iv. Oral Hygiene Index-Simplified (OHI-S): comprising Debris index (DI) and Calculus index (CI), each scored 0-3. OHI-S scored: good (0.0-1.2) to poor oral hygiene (3.1-6.0).

   v. Gingival index (GI): 0=normal gingiva, 3=severely inflamed gingiva/spontaneous bleeding.

   vi. Other lesions present (including HIV-associated oral lesions).

   Study Procedures/Data collection:

   One trained research assistant (RA) per site will be hired, trained, and calibrated (minimum kappa score: 0.8). Consented primary caregivers of eligible children will be contacted by RAs.

   Baseline data will be extracted from participants' clinic charts. OHRQoL will be assessed for each participant. Baseline oral health status will be assessed and scored per established guidelines following intra-oral clinical examination.

   All participants will be frequency matched.

   Intervention: Trained instructor will give 45-minute oral health education and instructions/training for self-oral care to groups of 4 or 5 children and primary caregivers along with cards for oral self care record purposes.

   The intervention will include oral hygiene instructions and motivation for oral self-care (dietary counseling; post-meal rinsing; flossing; brushing frequency, time, and method; tongue cleaning; toothbrush type/care; toothpaste quantity/type; dental visits). Audiovisual aids and leaflets reinforcing the oral health education will be provided. Reminders will be sent out monthly via text messages.

   Control arm: will not receive oral health intervention at the time of the study, but as soon as the period of the study is over, the intervention will be given.

   Participants with findings that require treatment will be linked to appropriate services and they will be financially responsible for such care. All participants will receive toothbrushes and toothpastes as incentive and funds for transportation cost during study visits.

   After baseline measurement and intervention to the intervention group, data collection for both groups will be done at 1 month, 3 months and 6, months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children aged 8-16 years (who can self-implement the oral health intervention with minimal caregiver supervision) attending selected clinics. HIV status will be based on clinic records.
* Primary caregiver consent; assent from child.
* On ART for ≥3 months.

Exclusion Criteria: Children who

* Have co-morbid conditions that increase their risk for oral diseases.
* Have good oral hygiene.
* Do not meet inclusion criteria.
* Decline assent or lack caregiver consent.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Oral Health Status | 6 months
  Oral Hygiene Index-Simplified (OHI-S) score
Gingival Health Status | 6 months
  Modified Gingival Index (MGI) score
Oral Health Related Quality of Life (OHRQoL) | 6 months
  Child Perception Questionnaire for varying ages 8 to 10 and 11 to 14 and upward (CPQ8-10, CPQ11-14)

SECONDARY OUTCOMES:
Dental Caries Status | One month
  Decayed, Missing, and Filled (DMFT/dmft) index
Dental Caries Sequelae | 6 months
  Pulp which is visible, Ulcerated oral mucosa, Fistula due to caries, Abscess due to caries (PUFA/pufa) index
Dental Caries Status | 6 months
  International Caries Detection and Assessment System (ICDAS)
HIV-associated oral lesions | One month
  Oral lesions that are associated with HIV
Other dental problems | One month
  Malocclusion, Molar-Incisor Hypomineralization (MIH), Trauma etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yewande I ADEYEMO, BDS, Principal Investigator — Bayero University, Kano/ Aminu Kano Teaching Hospital
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Nigeria

REFERENCES:
- [Derived] Adeyemo YI, Aliyu MH, Folayan MO, Coker MO, Riedy CA, Maiyaki BM, Denloye OO. A 2-arm randomized controlled study to improve the oral health of children living with HIV in Nigeria: Protocol and study design. Contemp Clin Trials. 2024 Jan;136:107375. doi: 10.1016/j.cct.2023.107375. Epub 2023 Oct 30. PMID 38404532